CLINICAL TRIAL: NCT03037437
Title: Modulation of Sorafenib Induced Autophagy Using Hydroxychloroquine in Hepatocellular Cancer
Brief Title: Sorafenib Induced Autophagy Using Hydroxychloroquine in Hepatocellular Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Sukeshi Patel, Principal Investigator, The University of Texas Health Science Center at San Antonio
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTMS 16-0076; HSC20160515H (Other: University of Texas Health Science Center- San Antonio)
Record Dates: First submitted 2017-01-19; First posted 2017-01-31 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2024-08

CONDITIONS: Hepatocellular Cancer
Keywords: Hepatocellular Cancer; Sorafenib; Hydroxychloroquine
MeSH Terms: conditions — Liver Neoplasms | interventions — Sorafenib; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- No prior systemic treatment (Experimental): Sorafenib (SOR)-naïve patients receive SOR 400 mg by PO twice daily on Cycle1/Day1 (C1D1). In clinical practice, dose reduction of SOR is often required. Therefore, on C1D15, the clinician will dose-reduce sorafenib based on toxicity and hydroxychloroquine (HCQ) 400 mg PO daily will be started. C2D1 of each cohort, toxicity of HCQ will be assessed. Dose reductions due to adverse events (AEs) to each agent are allowed for SOR per standard of care and/or HCQ for grade 3+ AE.
  Interventions: Drug: Sorafenib (SOR); Drug: Hydroxychloroquine (HCQ)
- Progress on sorafenib (Experimental): As second-line treatment, we will add hydroxychloroquine (HCQ) to sorafenib (SOR) dose the patient was tolerating at the time of progression.
  Interventions: Drug: Sorafenib (SOR); Drug: Hydroxychloroquine (HCQ)

INTERVENTIONS:
Drug: Sorafenib (SOR) — Patients will receive SOR 400 mg by PO twice daily on Cycle1/Day1 (C1D1).
  Other Names: Nexavar
Drug: Hydroxychloroquine (HCQ) — 400mg by mouth daily
  Other Names: Plaquenil

SUMMARY:
The PI is studying if sorafenib/hydroxychloroquine (HCQ) will have improved efficacy when compared to sorafenib alone and in patients progressing of sorafenib the addition of HCQ would lead to disease stability in patients with advanced hepatocellular cancer (HCC).

DETAILED DESCRIPTION:
Phase 2 study with two cohorts:

Cohort 1: As second-line treatment, we will add HCQ to SOR dose the patient was tolerating at the time of progression.

Cohort 2: SOR-naïve patients receive SOR 400 mg by PO twice daily on Cycle1 Day1 (C1D1). On Cycle 1 Day 15, HCQ 400 mg PO daily will be started. In clinical practice, dose reduction of SOR may be required. On C1D15 SOR maybe kept as starting dose or reduced for toxicity. On Cycle 2 Day 1 of toxicity of HCQ and SOR will be assessed.

Each cycle is 28 days.

Blood samples will be collected at Cycle 1 Day 1, Cycle 1 Day 15 and Cycle 2 Day 1 to assess for biomarkers.

Disease evaluation every 2 cycles.

Dose reductions due to adverse events are allowed for both sorafenib per standard of care and/or HCQ for grade 3 or more adverse event was related to study medication. Dose reductions are also permitted based on investigator clinical decision.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically confirmed advanced or metastatic HCC. If no histological diagnosis, patient must have imaging studies compatible with HCC.
* Age 18 years and above
* ECOG performance status of 0 or 1
* Not a candidate for curative treatments (i.e., resection, transplantation)
* Child-Pugh class A or B7 liver function
* Measurable disease as defined by RECIST 1.1
* Patients who received prior local therapy (e.g., TACE) are eligible.
* Documented virology status of hepatitis, as confirmed by screening HBsAg, anti-HBc, and/or anti-HCV
* Life expectancy> 3 months
* For women who are not postmenopausal (12 months of amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to use two adequate methods of contraception. For men: agreement to use a barrier method of contraception during the treatment period
* Hematologic, Biochemical, and Organ Function within 7 days prior to Cycle 1 Day 1: Granulocyte count > 1500/mm3, Platelet count > 75,000/ mm3, Hemoglobin > 8 g/dL; Total bilirubin < 2.0; Albumin > 2.8g/dl; AST (SGOT) and ALT (SGPT) < 5 x ULN; Serum creatinine< 1.5 x ULN
* Cohort 1 (with sorafenib): No previous systemic therapy including sorafenib or chemotherapy treatment. Previous TACE and local treatments are permitted.
* Cohort 2 (on progression of sorafenib): Patients who have received prior sorafenib therapy for at least 4 weeks and has confirmation of disease progression on CT/MRI. Prior surgery or local therapy within 4 weeks prior to Cycle 1 Day 1, with the exception of palliative radiation therapy to the bone

Exclusion Criteria:

* Patients receiving prior therapy with HCQ.
* Patients with uncontrolled brain metastases. Patients with brain metastases must be asymptomatic and off corticosteroids for at least one week.
* Due to risk of disease exacerbation, patients with psoriasis are ineligible unless the disease is well controlled, and they are under the care of a specialist for the disorder who agrees to monitor the patient for exacerbations.
* Patients with previously documented macular degeneration or or untreated diabetic retinopathy (stable retinopathy is allowed).
* Patients may not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to HCQ.
* Patients requiring the use of enzyme-inducing anti-epileptic medication (phenytoin, carbamazepine, phenobarbital, primidone or oxcarbazepine) are not eligible for entry into the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* QTc > 500 milliseconds (ms) at baseline.
* Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease. Patients with NG-tube, J-tube, or G-tube will not be allowed to participate.
* Pregnant women are excluded from this study because sorafenib has the potential for teratogenic or abortifacient effects. For this reason, women of childbearing potential and men must also agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation.
* Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with sorafenib, breastfeeding should be discontinued.
* Informed Consent - No study specific procedures will be performed without a written and signed informed consent document. Patients who do not demonstrate the ability to understand or the willingness to sign the written informed consent document will be excluded from study entry.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
Time to tumor progression evaluated via tumor imaging | Through study completion, an average of 1 year
  Computerized axial tomography (CAT) Scan or Magnetic resonance imaging (MRI) will be done at Screening, then every other cycle and evaluated using RECIST version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Sukeshi Patel Arora, MD, Principal Investigator — Cancer Therapy & Research Center University of Texas Health Science Center San Antonio
Locations (1):
- University of Texas Health Cancer Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No